CLINICAL TRIAL: NCT07197463
Title: Study on the Therapeutic Effect of Phase I Cardiac Rehabilitation on Elderly Patients With Coronary Heart Disease Complicated by Sarcopenia:A Single Center, Randomized Control Study in China
Brief Title: The Therapeutic Effect of Phase I Cardiac Rehabilitation on Elderly Patients With CHD Complicated by Sarcopenia
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Qilu Hospital of Shandong University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: KYLL-202504-007-1
Record Dates: First submitted 2025-07-25; First posted 2025-09-29 (Actual); Last update posted 2025-09-29 (Actual); Status verified 2025-09

CONDITIONS: Coronary Disease; Sarcopenia
MeSH Terms: conditions — Coronary Disease; Sarcopenia | interventions — Atorvastatin

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Phase I Cardiac Rehabilitation Experimental Group (Experimental): Phase I cardiac rehabilitation（ low-intensity resistance training, breathing exercises, and bedside cycling） + drug therapy （Aspirin, Atorvastatin, Nitroglycerin）+ general treatment（quit smoking）
  Interventions: Other: drug therapy （Aspirin, Atorvastatin, Nitroglycerin）+ general treatment（quit smoking）
- General Treatment Group (Active Comparator): drug therapy（Aspirin, Atorvastatin, Nitroglycerin）+ general treatment（quit smoking）
  Interventions: Other: drug therapy （Aspirin, Atorvastatin, Nitroglycerin）+ general treatment（quit smoking）

INTERVENTIONS:
Other: drug therapy （Aspirin, Atorvastatin, Nitroglycerin）+ general treatment（quit smoking） — The experimental group received Phase I cardiac rehabilitation intervention + medication treatment + general treatment, while the control group only received medication treatment + general treatment.

SUMMARY:
The purpose of this clinical trial is to explore whether Phase I cardiac rehabilitation can treat elderly patients with coronary heart disease complicated by sarcopenia. It will also investigate the mechanism of Phase I cardiac rehabilitation. The main questions it aims to answer are:

* Can Phase I cardiac rehabilitation enhance muscle strength ?
* Can Phase I cardiac rehabilitation reduce in vivo inflammatory indicators? Researchers will compare the experimental group (Phase I cardiac rehabilitation + drug therapy + general treatment) with the control group (drug therapy + general treatment) to see if Phase I cardiac rehabilitation can treat elderly patients with coronary heart disease complicated by sarcopenia and reduce inflammatory indicators.

Participants will:

* Receive Phase I cardiac rehabilitation training（mainly includes low-intensity resistance training, breathing training and bedside cycling） or conventional drug therapy for 3 consecutive months.
* Undergo examinations 10 days after training, 1 month after discharge, and 3 months after discharge respectively.
* Record changes in their muscle strength and blood inflammatory indicators.

DETAILED DESCRIPTION:
The main purpose of this study is to explore the clinical efficacy of Phase I cardiac rehabilitation in the treatment of elderly patients with coronary heart disease complicated by sarcopenia and its potential clinical mechanisms.

The determination of this sample size is based on research hypotheses and estimates of the expected efficacy level, calculated in accordance with statistical principles. The PASS software was used for sample size estimation, with a significance level (alpha) of 0.050. Using the two independent samples t-test, 15 cases in the experimental group and 15 cases in the control group were needed to achieve a test power of >90%. To enhance the statistical power of the results, it was decided to include 50 cases in the experimental group and 50 cases in the control group, totaling 100 patients.

Research participants with high compliance were screened. Before the start of the clinical trial, researchers provided sufficient education to the participants, including the trial process, potential benefits and risks, as well as the rights and obligations of the participants. Only after the participants fully understood the trial and signed the informed consent form could they be enrolled.

SPSS generated a random number table. According to the table, odd numbers were assigned to the intervention group and even numbers to the control group, and simple randomization was used for group allocation. Statistical result analysis will be conducted at the 0.05 significance level, using SPSS statistical software.

Risk monitoring will be carried out during the trial: closely observe abnormal situations during the trial to prevent risks; promptly identify various types of risks; and on the basis of risk identification, conduct risk assessment. If risks occur, corresponding risk handling strategies will be formulated according to different risk levels. In the event of a serious adverse event, researchers will report it to the regulatory authorities and the ethics committee within 24 hours and fill out a serious adverse event report form.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 60 years;
* Coronary heart disease confirmed by coronary CTA or coronary angiography, with stable condition within the past 8 hours, including: ① no new or recurrent chest pain; ② no further elevation of troponin level; ③ no new signs of decompensated heart failure (dyspnea at rest accompanied by moist rales); ④ no new malignant arrhythmias or dynamic changes in electrocardiogram. Basic vital signs are normal, including: ① resting heart rate of 50-100 beats per minute; ② resting blood pressure of 90-150/60-100 mmHg (1 mmHg = 0.133 kPa); ③ oxygen saturation > 95%.
* Meeting the diagnostic criteria for sarcopenia (2024 Edition of Chinese Guidelines for the Diagnosis and Treatment of Sarcopenia);
* Having good compliance to ensure the completion of this study;
* Being able to understand the purpose of the trial, voluntarily participating in the study and signing the informed consent form.

Exclusion Criteria:

* Severe arrhythmia, decompensated heart failure, severe respiratory failure, untreated severe aortic stenosis, acute aortic dissection, resting hypertension with systolic and/or diastolic blood pressure > 200/110 mmHg;
* Mental disorders with limited cooperation ability; severe cognitive or behavioral disorders; end-stage diseases; acute diseases (e.g., acute infections, injuries) that restrict physical activity;
* Poor compliance and inability to cooperate with the completion of this study.

Ages: 60 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2025-10-10 (Estimated); Primary Completion 2026-10-10 (Estimated); Study Completion 2026-11-10 (Estimated)

PRIMARY OUTCOMES:
Change in Grip Strength | From enrollment（ baseline）to 1 month after treatment initiation
  The primary outcome measure is the change in muscle strength.Muscle strength is measured using a hand dynamometer. Participants are instructed to grip the dynamometer with their dominant hand at maximum effort, and the maximum grip force value is recorded (unit: kgf).

SECONDARY OUTCOMES:
Change in Grip Strength | From enrollment（ baseline）to 3 month after treatment initiation
  The primary outcome measure is the change in muscle strength.Muscle strength is measured using a hand dynamometer. Participants are instructed to grip the dynamometer with their dominant hand at maximum effort, and the maximum grip force value is recorded (unit: kgf).

CONTACTS AND LOCATIONS:
Overall Officials: Yanyan Hu, Doctor, Study Chair — Qilu Hospital of Shandong University

IPD SHARING:
Plan to Share IPD: No